CLINICAL TRIAL: NCT02526342
Title: Impact of Negative Pressure Wound Therapy on Free Muscle Flaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulf Dornseifer, MD (Other)
Responsible Party: Sponsor-Investigator, Ulf Dornseifer, MD, Dr.med., Klinik Bogenhausen
Organization: Klinik Bogenhausen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBogenhausen_04
Record Dates: First submitted 2015-08-02; First posted 2015-08-18 (Estimated); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Negative-Pressure Wound Therapy; Edema; Free Flap; Microcirculation; Macrocirculation
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Negative Pressure Wound Therapy (Active Comparator): Patients receive a Negative Pressure Wound Therapy-Dressing (V.A.C. Ultra (KCI®,San Antonio, Texas, USA) with a subatmospheric pressure of 125mmHg to cover the muscle flap for five days following surgery.
  Interventions: Device: V.A.C. UltraTM (KCI®,San Antonio, Texas, USA)
- Conventional Dressing (No Intervention): Patients receive a conventional dressing for the muscle flap including fatty gauze and cotton gauze.

INTERVENTIONS:
Device: V.A.C. UltraTM (KCI®,San Antonio, Texas, USA) — Free muscle flaps are treated with Negative Pressure Wound Therapy (V.A.C. Ultra (KCI®,San Antonio, Texas, USA)) for five days following surgery with a continuous subatmospheric pressure of 125 mmHg.
  Arms: Negative Pressure Wound Therapy

SUMMARY:
Aim of the study is to prove the utility and safety of the negative pressure wound therapy (NPWT) in the postoperative management of free flaps.

The quantitative assessment of the entirety of clinical main relevant parameters like edema formation, microcirculation, macrocirculation and wound healing should create a better and comprehensive understanding of the NPWT effects in this field.

DETAILED DESCRIPTION:
This study evaluates the impact of negative pressure wound therapy on free muscle flaps. Flaps were treated with NPWT or with a conventional dressing (control) for five days following tissue transfer. Edema formation is measured by a 3D scan (Artec SpiderTM) during the operation, five and fourteen days after surgery. The macrocirculation- and microcirculation parameters of the flaps are assessed using an implanted Doppler probe (Cook-Swartz®) as well as combined flowmetry and remission spectroscopy (O2C®). These measurements are conducted daily at the day of the operation as well as the first five days following the operation. Following dressing removal at the fifth postoperative day, skin graft take is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring free muscle flap reconstruction at the lower extremity covered with a split thickness skin graft
* existing cognitive faculty
* consent

Exclusion Criteria:

* non-compliance
* non-consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-07-18 (Actual); Study Completion 2016-07-18 (Actual)

PRIMARY OUTCOMES:
Change of Flap Edema in the early postoperative period measured by a 3D Scan - Artec SpiderTM, Artec Group, Palo Alto, California, USA | Measurements were conducted at the day of the operation, five and fourteen days following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Dornseifer, M.D., Principal Investigator — Bogenhausen Academic Hospital, Technische Universität München, Munich, Germany
Locations (1):
- Department of Plastic, Reconstructive, Hand and Burn Surgery, Bogenhausen Academic Hospital, Technische Universität München, Munich, Germany